CLINICAL TRIAL: NCT05825235
Title: Long-term Efficacy and Tolerability of add-on Pramipexole for Anhedonic Depression - an Open Label Follow-up Study
Brief Title: Long-term Efficacy of Pramipexole in Anhedonic Depression
Acronym: LONG-PRAXOL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-502270-17-00
Record Dates: First submitted 2023-03-23; First posted 2023-04-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Anhedonia; Depression
Keywords: anhedonia; depression; dopamine; pramipexole
MeSH Terms: conditions — Anhedonia; Depression | interventions — Pramipexole

STUDY DESIGN:
Intervention Model Description: Within the frame of the previous RCT study (Eudra CT 2022-001563-26) approximately 50% of the participants have been treated with the study product and 50% with placebo. In this study all participants receive the study product, so some will continue their ongoing treatment with the study product and some will start using the study product.
Masking Description: Not masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pramipexole (Experimental): Pramipexole prolonged-release tablet with doses ranging from 0.26 mg base to 3.15 mg base / day, study duration 6 months
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Pramipexole — 6 months of treatment with add-on Pramipexole

SUMMARY:
The purpose of the study is to assess the long-term efficacy and safety of add-on pramipexole for treatment of patients with anhedonic depression.

DETAILED DESCRIPTION:
The heterogeneity of depression suggests that several different neurocircuits and pathophysiological mechanisms are involved. Anhedonia - the inability to experience pleasure from, or the lack of motivation to carry out, usually enjoyable activities - is a promising endophenotype within the depression spectrum, with a distinct pathophysiology involving dopaminergic mesolimbic projections. Anhedonia is common in depression and associated with treatment resistance. Pramipexole, an agonist to the dopamine -receptor 3, is an established treatment of Parkinson's disease. Based on its mechanism of action, pramipexole might be efficacious in a subtype of depression characterized by anhedonia and lack of motivation - symptoms linked to dopaminergic hypofunction.

The aim of this open label follow-up study is to test the long-term efficacy and tolerability of add-on pramipexole in anhedonic depression. This is a continuation study of an RCT (EudraCT# 2022-001563-26) in which patients are randomized to either pramipexole or placebo for 9 weeks. After completion of the RCT, patients will be offered to participate in the current trial. Approximately 50% of the patients have been treated with pramipexole and 50% with placebo within the frames of the RCT. Patients randomized to pramipexole in the RCT will continue on their current dose and patients randomized to placebo will start pramipexole using the same dosing schedule as in the RCT. A total of 80 research subjects with unipolar depression, bipolar disorder in depressive phase, or dysthymia will be offered participation in the study after completing the RCT given that they fulfill all the inclusion criteria, and none of the exclusion criteria.

Subjects have study visits once a month during 6 months, or more often if needed based on side effects. Symptom severity, side effects and ecological momentary assessments are recorded at each study visit and dose titration schedule is modified as needed. Between study visits, research subjects may contact study personnel and the investigators can quickly arrange for an additional study visit if needed.

After the study, the decision to continue with pramipexole outside of the study or discontinue with pramipexole will be based on patient preference in combination with a willingness of the patient's regular physician to take over the treatment outside of the study.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in RCT testing the short-term efficacy of pramipexole vs placebo (EudraCT# 2022-001563-26).
* Study participants randomized to pramipexole in the RCT who wish to continue with their treatment can enrol in the study.
* Study participants randomized to placebo in the RCT who continue to fulfil the inclusion criteria (and none of the exclusion criteria) after the RCT can enrol in the study.
* The research subject has given informed consent to participate in the study.

Additional inclusion criterion for patients receiving placebo during the RCT

* Anhedonia symptoms: 3 or 4 points on ≥ 3 items of the Snaith-Hamilton Pleasure Scale (SHAPS-C). This has been adopted in previous studies as a definition of "clinically significant anhedonia".

Exclusion Criteria:

* Pregnancy, breastfeeding or planned pregnancy (if female).
* High suicide risk according to the overall clinical assessment of the research physician.
* Ongoing substance abuse (within 6 months).
* Diagnosis of current psychosis.
* Known diagnosis of Emotionally Unstable Personality Disorder.
* Treatment under LPT.
* History of impulse control disorder (including current binge-eating disorder) or a current ADHD diagnosis with hyperactivity.
* Diagnosis of intellectual disability, dementia, or other circumstance that makes it difficult to understand the meaning of participating in the trial and give informed consent.
* Diagnosis of renal failure or severe cardiovascular disease (specifically symptomatic heart failure NYHA Class II). Blood samples from RCT are sufficient to rule this out.
* Recently started psychotherapy (within 6 weeks) or planning to start such treatment during participation in the trial.
* Ongoing ECT, ketamine or rTMS treatment, excluding maintenance ECT, ketamine or rTMS (Maintenance treatment is defined as the use of ECT/ketamine/rTMS for a period exceeding 3 months after a series of ECT/ketamine/rTMS treatment in order to prevent the onset of a new episode).
* Other medical conditions or other concomitant drug treatment (see section 14.5) which, in the opinion of the investigators, may affect the evaluability of the trial or conditions that increase trial risk. For example, Parkinson's disease, hepatic insufficiency, ongoing cancer not in remission for more than one year, gastric bypass surgery that affects the absorption of extended release tablets.
* Known or suspected allergy to any active substance or excipient in the medicinal product included in the trial.
* Participation in other treatment studies.
* Other reason, as assessed by the investigator, that prevents the research subject's participation, such as the risk that the research subject is unable to complete the trial (non-compliance).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Anhedonia symptoms | Baseline
  Total Snaith Hamilton Anhedonia Pleasure (SHAPS) self-report scale scores. Higher scores equal more severe anhedonoa. Score range 14-56
Anhedonia symptoms | Month 1
  Total SHAPS self-report scores. Higher scores equal more severe anhedonoa. Score range 14-56
Anhedonia symptoms | Month 2
  Total SHAPS self-report scores. Higher scores equal more severe anhedonoa. Score range 14-56
Anhedonia symptoms | Month 3
  Total SHAPS self-report scores. Higher scores equal more severe anhedonoa. Score range 14-56
Anhedonia symptoms | Month 4
  Total SHAPS self-report scores. Higher scores equal more severe anhedonoa. Score range 14-56
Anhedonia symptoms | Month 5
  Total SHAPS self-report scores. Higher scores equal more severe anhedonoa. Score range 14-56
Anhedonia symptoms | Month 6
  Total SHAPS self-report scores. Higher scores equal more severe anhedonoa. Score range 14-56

SECONDARY OUTCOMES:
Core depression symptoms | baseline
  Hamilton Depression Rating Scale-6 (HDRS6) scores (subscale of HDRS-17)
Core depression symptoms | Month 1
  HDRS6 scores (subscale of HDRS-17)
Core depression symptoms | Month 2
  HDRS6 scores (subscale of HDRS-17)
Core depression symptoms | Month 3
  HDRS6 scores (subscale of HDRS-17)
Core depression symptoms | Month 4
  HDRS6 scores (subscale of HDRS-17)
Core depression symptoms | Month 5
  HDRS6 scores (subscale of HDRS-17)
Core depression symptoms | Month 6
  HDRS6 scores (subscale of HDRS-17)
Ecological momentary assessments | baseline
  Number of steps/day, movement pattern distribution over the day, walking distance, time spent in light, moderate and intense physical activity, resting heart rate, blood oxygen saturation, heart rate variability (stress scores), sleep latency (time to fall asleep), sleep awakening (how often you wake up during the night), wakefulness (time in minutes awake during a night), time in deep sleep, sleep efficiency (time asleep vs. total time in bed). All variables are measured using activity meters.
Ecological momentary assessments | Month 1
  By using activity meters, we will analyze relevant outcomes related to physical activity, sleep, and heart rate
Ecological momentary assessments | Month 2
  By using activity meters, we will analyze relevant outcomes related to physical activity, sleep, and heart rate
Ecological momentary assessments | Month 3
  By using activity meters, we will analyze relevant outcomes related to physical activity, sleep, and heart rate
Ecological momentary assessments | Month 4
  By using activity meters, we will analyze relevant outcomes related to physical activity, sleep, and heart rate
Ecological momentary assessments | Month 5
  By using activity meters, we will analyze relevant outcomes related to physical activity, sleep, and heart rate
Ecological momentary assessments | Month 6
  By using activity meters, we will analyze relevant outcomes related to physical activity, sleep, and heart rate
Anhedonic symptoms | baseline
  Dimensional Anhedonia Rating Scale (DARS) total score
Anhedonic symptoms | Month 1
  Dimensional Anhedonia Rating Scale (DARS) total score
Anhedonic symptoms | Month 2
  Dimensional Anhedonia Rating Scale (DARS) total score
Anhedonic symptoms | Month 3
  Dimensional Anhedonia Rating Scale (DARS) total score
Anhedonic symptoms | Month 4
  Dimensional Anhedonia Rating Scale (DARS) total score
Anhedonic symptoms | Month 5
  Dimensional Anhedonia Rating Scale (DARS) total score
Anhedonic symptoms | Month 6
  Dimensional Anhedonia Rating Scale (DARS) total score
General depressive symptoms | baseline
  Montgomery-Åsberg Depression Rating Scale (MADRS-S)
General depressive symptoms | Month 1
  Montgomery-Åsberg Depression Rating Scale (MADRS-S)
General depressive symptoms | Month 2
  Montgomery-Åsberg Depression Rating Scale (MADRS-S)
General depressive symptoms | Month 3
  Montgomery-Åsberg Depression Rating Scale (MADRS-S)
General depressive symptoms | Month 4
  Montgomery-Åsberg Depression Rating Scale (MADRS-S)
General depressive symptoms | Month 5
  Montgomery-Åsberg Depression Rating Scale (MADRS-S)
General depressive symptoms | Month 6
  Montgomery-Åsberg Depression Rating Scale (MADRS-S)
Sleep and insomnia | Baseline
  Insomnia Severity Index (ISI) total score
Sleep and insomnia | Month 1
  Insomnia Severity Index (ISI) total score
Sleep and insomnia | Month 2
  Insomnia Severity Index (ISI) total score
Sleep and insomnia | Month 3
  Insomnia Severity Index (ISI) total score
Sleep and insomnia | Month 4
  Insomnia Severity Index (ISI) total score
Sleep and insomnia | Month 5
  Insomnia Severity Index (ISI) total score
Sleep and insomnia | Month 6
  Insomnia Severity Index (ISI) total score
Apathy symptoms | Baseline
  Apathy Evaluation Scale (AES) total score
Apathy symptoms | Month 1
  Apathy Evaluation Scale (AES) total score
Apathy symptoms | Month 2
  Apathy Evaluation Scale (AES) total score
Apathy symptoms | Month 3
  Apathy Evaluation Scale (AES) total score
Apathy symptoms | Month 4
  Apathy Evaluation Scale (AES) total score
Apathy symptoms | Month 5
  Apathy Evaluation Scale (AES) total score
Apathy symptoms | Month 6
  Apathy Evaluation Scale (AES) total score
Anxiety symptoms | baseline
  Generalized Anxiety Disorder 7-item scale (GAD-7)
Anxiety symptoms | Month 1
  Generalized Anxiety Disorder 7-item scale (GAD-7)
Anxiety symptoms | Month 2
  Generalized Anxiety Disorder 7-item scale (GAD-7)
Anxiety symptoms | Month 3
  Generalized Anxiety Disorder 7-item scale (GAD-7)
Anxiety symptoms | Month 4
  Generalized Anxiety Disorder 7-item scale (GAD-7)
Anxiety symptoms | Month 5
  Generalized Anxiety Disorder 7-item scale (GAD-7)
Anxiety symptoms | Month 6
  Generalized Anxiety Disorder 7-item scale (GAD-7)
Life quality | Baseline
  Brunnsviken Brief Quality of life scale (BBQ) total score
Life quality | Month 1
  Brunnsviken Brief Quality of life scale (BBQ) total score
Life quality | Month 2
  Brunnsviken Brief Quality of life scale (BBQ) total score
Life quality | Month 3
  Brunnsviken Brief Quality of life scale (BBQ) total score
Life quality | Month 4
  Brunnsviken Brief Quality of life scale (BBQ) total score
Life quality | Month 5
  Brunnsviken Brief Quality of life scale (BBQ) total score
Life quality | Month 6
  Brunnsviken Brief Quality of life scale (BBQ) total score
Side effects | Baseline
  Number and severity of adverse events
Side effects | Month 1
  Number and severity of adverse events
Side effects | Month 2
  Number and severity of adverse events
Side effects | Month 3
  Number and severity of adverse events
Side effects | Month 4
  Number and severity of adverse events
Side effects | Month 5
  Number and severity of adverse events
Side effects | Month 6
  Number and severity of adverse events
Cognitive symptoms | 6 months
  Change in cognitive performance using the WAIS-IV, Repeatable Battery for the Assessment of Neuropsychological Status, Delis-Kaplan Executive Function System.

CONTACTS AND LOCATIONS:
Locations (1):
- Region Skåne, Lund, Skåne County, Sweden

REFERENCES:
- [Derived] Lindahl J, Asp M, Stahl D, Tjernberg J, Eklund M, Bjorkstrand J, van Westen D, Jensen J, Mansson K, Tornberg A, Svensson M, Deierborg T, Ventorp F, Lindqvist D. Add-on pramipexole for anhedonic depression: study protocol for a randomised controlled trial and open-label follow-up in Lund, Sweden. BMJ Open. 2023 Nov 30;13(11):e076900. doi: 10.1136/bmjopen-2023-076900. PMID 38035737